CLINICAL TRIAL: NCT00242294
Title: A Confirmatory Study of APTA-2217 in Patients With Chronic Obstructive Pulmonary Disease (A Placebo-controlled Double-blind Comparative Study)
Brief Title: Efficacy and Safety of Roflumilast in Japanese Patients Older Than 40 Years With Chronic Obstructive Pulmonary Disease (APTA-2217-06)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APTA-2217-06
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Phosphodiesterase 4 inhibitor; Roflumilast
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

INTERVENTIONS:
Drug: Roflumilast

SUMMARY:
The aim of the study is to investigate the effect of roflumilast (APTA-2217) on lung function in patients with chronic obstructive pulmonary disease (COPD). Roflumilast will be administered orally once daily. The study duration consists of a baseline period (4 weeks) and a treatment period (24 weeks). The study will provide further data on safety, tolerability, and effectiveness of roflumilast.

ELIGIBILITY:
Main inclusion criteria:

* Patients with chronic obstructive pulmonary disease
* Current smoker or ex-smoker
* 30 to 80% of predicted FEV1 after inhalation of short acting beta stimulant

Main exclusion criteria:

* Patients with poorly controlled COPD
* Patients who need for long-term oxygen therapy
* Patients who have concurrent respiratory diseases such as asthma, diffuse panbronchiolitis, congenital sinobronchial syndrome, bronchiolitis obliterans, bronchiectasis, active tuberculosis, pneumoconiosis, pulmonary lymph vascular myoma, which are considered to affect the evaluation

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 570
Dates: Start 2004-11; Primary Completion 2006-09 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
change in lung function parameters (post-bronchodilator).

SECONDARY OUTCOMES:
pulmonary function test, COPD symptoms, rescue medication, evaluation of QOL, COPD exacerbation, adverse events, pharmacokinetics.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Nycomed Japan and Mitsubishi Tanabe Oharma Corporation, Osaka, Japan

REFERENCES:
- See also: APTA-2217-06-RDS-2008-12-05.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4466&filename=APTA-2217-06-RDS-2008-12-05.pdf